CLINICAL TRIAL: NCT03036228
Title: MTH1, A Phase I, Study on Tumors Inhibition, First in Human, First in Class
Acronym: MASTIFF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Helleday Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MASTIFF
Record Dates: First submitted 2017-01-13; First posted 2017-01-30 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Solid tumours
MeSH Terms: conditions — Neoplasms | interventions — karonudib

STUDY DESIGN:
Intervention Model Description: First part of the study - different dose cohorts with escalating doses. Extension part - Characterization of the Phase 2 Recommended Dose (P2RD) in specific patient groups and correlation with clinical outcome and other PD markers is currently examined.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation (Experimental): Karonudib is an oral inhibitor of MTH1 supplied as an oral solution and now as tablets. Each cycle is defined as 28 days.
  Interventions: Drug: Karonudib

INTERVENTIONS:
Drug: Karonudib — Dose escalation of administration with Karonudib.

SUMMARY:
Primary Objective

• To determine the safety and tolerability of Karonudib (TH1579) in escalating doses for the treatment of patients with advanced solid malignant tumours.

Secondary Objective

* To define DLT and MTD.
* To determine a recommended phase 2 dose (RP2D) and schedule.
* To determine the pharmacokinetics of Karonudib.
* To determine preliminary signs of clinical efficacy of Karonudib.
* To determine overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age at least 18 years (there is no upper age limit but patients must be judged to have a "biologic" age of 75 years or less).
3. Life expectancy of at least 12 weeks (as per investigators clinical assessment).
4. ECOG PFS 0 or 1.
5. Patients must have measurable disease based on RECIST 1.1 criteria or evaluable metastatic disease unless otherwise specified in specific patient groups.
6. Patients with any 1 of the following histologically confirmed tumors and who qualifies for new therapy and relapsing to/after standard therapy or the patient has refused or does not tolerate standard therapy Cohort 19

   1. Histologically or cytologically confirmed adenocarcinoma of prostate that is metastatic, hormone-refractory (confirmed by testing serum testosterone), and clinically progressive following at least one prior hormonal regimen. Prostate cancer patients must have measurable (patient with measurable bi-dimensional disease) or evaluable disease (defined as the presence of a non-measurable abnormality on CT or on physical examination coupled with an abnormal PSA value) or PSA relapse (Obtain sequence of rising values at a minimum of 1-week intervals, 1.0 ng/mL minimal value). Patients can only have received a taxane therapy in the pre-metastatic hormone refractory setting
   2. High Grade Serous Ovarian, Fallopian Tube or Primary Peritoneal Cancer that can be assessed radiological, clinically or biochemically.
   3. Cytologically or histologically confirmed endometrial cancer that is recurrent or metastatic and/or resistant to standard therapies, or for which no standard therapy is available. Patients must have measurable disease based on RECIST 1.1 criteria or evaluable metastatic disease.

      Cohort 20
   4. Biopsy-proven carcinoma of the cervix that is either locally advanced or metastatic.
   5. Recurrent or metastatic head and neck adenocarcinoma who are not candidates for curative surgery or refusing surgical treatment
7. Adequate bone marrow, hepatic and renal function defined as:

   1. Haemoglobin ≥ 95 g/L (blood transfusion not less than 21 days prior to screening).
   2. Absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥100 x 109/L.
   3. Total bilirubin < 1.5 x ULN (does not apply to patients with Gilberts Syndrome).
   4. AST and ALT ≤ 1.5 x ULN (or ≤ 3 x ULN in the presence of liver metastases).
   5. Serum creatinine not over ≤ ULN (if serum creatinine is between 1 and 1.5 x ULN, patients may be eligible provided that the calculated GFR is at least 50 ml/min using Cockcroft-Gault method).
   6. Albumin greater than or equal to 23 g/L.
8. Subject must be able to take oral medication.
9. Negative pregnancy test according to CTFG guidance 2014 for females of child-producing potential.
10. Known HIV-infected patients with undetectable viral loads will be eligible for the study. HIV testing is mandatory

Exclusion Criteria:

1. Age less than 18 years.
2. Less than 4 weeks since stopping previous systemic cancer treatment or less than 5 half lifes of prior therapy, whichever is shorter.
3. Less than 3 weeks since stopping palliative radiotherapy.
4. Less than 3 weeks after minor surgery.
5. Less than 6 months since a clinically significant cardiovascular event such as myocardial infarction, unstable angina, angioplasty, bypass surgery, stroke or TIA.
6. Congestive heart failure NYHA class ≥ II.
7. History of arrhythmias or arrhythmias discovered during the screening period (apart from atrial fibrillation without ventricular tachycardia and premature extra beats).
8. Patients requiring anti-arrhythmic drugs.
9. QTc interval >450 ms at baseline.
10. Use of fentanyl (must be stopped at least 1 week prior to initiation of Karonudib).
11. Use of anti-oxidants vitamins and acetylcysteine (must be stopped within 48 hours of starting treatment with Karonudib).
12. Use of antidepressant medications which are substrate for CYP2D6 (must be stopped at least 3 weeks prior to starting treatment with Karonudib).
13. Any severe acute or chronic medical condition that places the patient at increased risk or interferes with the interpretation of study results.
14. Leptomeningeal metastases (patient with previously treated brain metastases are eligible provided that there is no evidence of disease progression for a minimum of 8 weeks prior to inclusion - in these cases a CNS MR is required within the screening period).
15. Known acute or chronic infection with hepatitis B or C that is untreated.
16. Pregnant or breast-feeding women.
17. Patients with reproductive potential not implementing accepted and effective means of contraception.
18. Participation in any other clinical trial within the previous 4 weeks.
19. Unable to comply with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Karonudib (TH1579) will be evaluated. | 28 days, first treatment cycle for the patient.
  Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD). DLTs will be assessed during first cycle of therapy, week 1-4 based on Haematological toxicity and Non-haematological toxicity.
  MTD: The highest dose of Karonudib that does not cause unacceptable side effects is defined as the MTD.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of Karonudib. | 28 days, first treatment cycle for the patient
  Peak Plasma Concentration, Cmax
To determine the pharmacokinetics of Karonudib. | 28 days, first treatment cycle for the patient
  Tmax, time is the time to reach Cmax (Peak Plasma Concentration)
To determine the pharmacokinetics of Karonudib. | 28 days, first treatment cycle for the patient
  biological half-life (plasma T1/2)
To determine the pharmacokinetics of Karonudib. | 28 days, first treatment cycle for the patient
  Area under the Curve (AUC)
To determine preliminary signs of clinical efficacy of Karonudib. | 54 days, two treatment cycles for the patient
  RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, BSc, Study Director — Oxcia
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala